CLINICAL TRIAL: NCT02522091
Title: Cerebral Substrates of Prospective Memory in Young and Its Disruption in Normal Aging and in Alzheimer's Disease: A Study in Anatomical MRI, Diffusion Tensor MRI and Functional MRI
Acronym: IMPRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10-002
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- young healthy volunteers (18-44 years old) (Other): young healthy volunteers (18-44 years old)
  Interventions: Device: functional brain MRI; Other: Neuropsychology tests
- healthy volunteers (45-69 years old) (Other): healthy volunteers (45-69 years old)
  Interventions: Device: functional brain MRI; Other: Neuropsychology tests
- Mild Cognitive Impairment Patients (Other): Mild Cognitive Impairment Patients
  Interventions: Device: functional brain MRI; Other: Neuropsychology tests
- Alzheimer's Disease patient (Other): Alzheimer's Disease patient
  Interventions: Device: functional brain MRI; Other: Neuropsychology tests
- old healthy volunteers (70+ years old) (Other): old healthy volunteers (70+ years old)
  Interventions: Device: functional brain MRI; Other: Neuropsychology tests

INTERVENTIONS:
Device: functional brain MRI
Other: Neuropsychology tests

SUMMARY:
Investigators propose in this study to evaluate prospective memory (MP) in all its complexity as well as the processes, cognitive and brain, the underlying. Specifically, investigators propose to evaluate the evolution of the MP during normal aging and Alzheimer's disease (AD) to identify the cognitive and brain processes underlying this development. To do this, this study will have to include healthy subjects, 18 to 95 years, patients with Mild Cognitive Impairment (MCI) and patients with probable AD. All participants will undergo a series of examinations, both neuropsychological and brain imaging.

ELIGIBILITY:
Inclusion Criteria:

* All participants:

  * Normal Education> 7 years
  * French mother tongue
  * right-handed (Edinburgh Inventory)
  * score on the scale of Beck <7 (depression scale)
  * signing the informed consent of the protocol in agreement with the Committee to Protect People
  * Medical examinations, neurological, neuropsychological and neuroimaging depth in accordance with the specific inclusion and exclusion criteria for each population, that is to say:
* Young healthy subjects aged between 18 and 44 years
* Healthy subjects intermediate age: between 45 and 69 years

  * score on the Mattis Dementia Scale higher than 137, in order to exclude any potential dementia
  * Performance "normal" to test RI RL-16 (that is to say, not differing by more than 1.65 standard deviation from the norm for age and cultural level [see normative values published Van der Linden et al., 2004]), test conventionally used to assess the verbal episodic memory.
* Healthy elderly subjects aged 70 and over, living at home

  * score on the Mattis Dementia Scale higher than 137, in order to exclude any potential dementia
  * Performance "normal" to test RI RL-16 (that is to say, not differing by more than 1.65 standard deviation from the norm for age and cultural level [see normative values published Van der Linden et al., 2004]), test conventionally used to assess the verbal episodic memory.
* MCI patients: older than 50 years and recruited from memory clinics and meet the current criteria and recognized including amnestic MCI

  * memory complaint
  * targets deficits of episodic memory (lower performance of at least 1 standard deviation from the norm for age and cultural level to one or more (sub) episodic memory scores of diagnostic battery - cf. . Tables 1 and infra)
  * performance in the standards for age and cultural level in all tests of diagnostic battery measuring other cognitive functions as memory, including the evaluation of overall cognitive ability tests.
* Alzheimer's patients: older than 50 years were recruited from the clinics and memory satisfying the standards NINCDS-ADRDA criteria for probable AD which include

  * abnormal global cognitive functioning and deficits in two or more cognitive domains identified by the diagnostic battery
  * mild to moderate AD (MMSE ≥ 18).

Exclusion Criteria:

* Cognitive disorders of sudden onset (contrary to their slow and progressive onset in AD), which could reflect a stroke; a modified Hachinski ischemic score ≤ 2 (Loeb & Gandolfo, 1983); history of head trauma with loss of consciousness for more than 1 hour, or encephalitis;
* Chronic neurological disease, psychiatric, endocrine, hepatic, infectious;
* A history of major illness (chronic lung disease, heart disorder, metabolic, hematologic, endocrine or immunological severe, cancer);
* A medication that may interfere with the mnemonic or metabolic measures (psychotropics, hypnotics, anxiolytics, neuroleptics, anti-Parkinson, benzodiazepines, anti-inflammatory drugs, antiepileptics, antihistamines, analgesics and muscle relaxants central, as is usual The investigating doctor deems the annoying character for the study of the regular intake of certain medications). Taking anticholinesterase treatment will also be a criterion for non-inclusion.
* Chronic intake of alcohol or drugs;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2010-11; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
measuring the amplitude of the BOLD signal (Blood Oxygen Level Dependent) | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Service de neurologie, Caen, CHU, France